CLINICAL TRIAL: NCT00190541
Title: Mesorectal Excision With Lateral Lymph Node Dissection Versus Without Lateral Lymph Node Dissection for Clinical Stage II, III Lower Rectal Cancer (JCOG0212)
Brief Title: Mesorectal Excision (ME) Versus ME With Lateral Node Dissection for Stage II, III Lower Rectal Cancer (JCOG0212)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Haruhiko Fukuda (Other)
Collaborators: Ministry of Health, Labour and Welfare, Japan (Other Government)
Responsible Party: Sponsor-Investigator, Haruhiko Fukuda, JCOG Data Center, Japan Clinical Oncology Group
Organization: Japan Clinical Oncology Group (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JCOG0212; C000000034 (Registry Identifier: UMIN-CTR)
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Last update posted 2016-09-22 (Estimated); Status verified 2016-09

CONDITIONS: Rectal Neoplasms
Keywords: Rectal Cancer; Lymph Node Dissection; Rectal Surgery; Autonomic Nerves; Stage II, III lower rectal cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Procedure/Surgery: Mesorectal excision with lateral lymph node dissection
  Interventions: Procedure: Mesorectal excision with lateral lymph node dissection
- 2 (Experimental): Procedure/Surgery: Mesorectal excision without lateral lymph node excision
  Interventions: Procedure: Mesorectal excision without lateral lymph node excision

INTERVENTIONS:
Procedure: Mesorectal excision with lateral lymph node dissection — Mesorectal excision with lateral lymph node dissection
  Arms: 1
Procedure: Mesorectal excision without lateral lymph node excision — Mesorectal excision without lateral lymph node excision
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the of international standard operation, mesorectal excision (ME alone) compared to Japanese standard operation, ME with lateral lymph node dissection for clinical stage II, III lower rectal cancer

DETAILED DESCRIPTION:
Total mesorectal excision (TME) or mesorectal excision (ME) with lateral lymph node dissection for advanced rectal cancer is widely performed in Japan. In other countries, TME or ME without lateral lymph node dissection is the standard. In order to determine which is the better rectal cancer surgery, relapse-free survivals of these are compared as the primary endpoint.

ELIGIBILITY:
Inclusion Criteria:

Preoperative criteria:

1. Histologically confirmed adenocarcinoma
2. Clinical stage II or III
3. Preoperative findings:

   * Main lesion of the tumor is located at the rectum
   * Lower tumor margin is below the peritoneal reflection
   * No extramesorectal lymph node swelling (Shorter diameter is less than 10 mm)
   * No invasion to other organ (s)
4. Patient age is more than 20 and less than 75
5. PS: 0, 1
6. No past history of chemotherapy, pelvic surgery or radiation
7. Written informed consent

   Operative criteria:
8. Mesorectal excision is performed
9. Operative findings:

   * Main lesion of the tumor is located at the rectum
   * Lower tumor margin is below the peritoneal reflection
10. R0 after resection

Exclusion Criteria:

1. Multiple cancer patients
2. Pregnant patients
3. Psychological disorder
4. Steroid administration
5. Cardiac infarction within six months
6. Severe pulmonary emphysema and pulmonary fibrosis
7. Doctor's decision for exclusion

Ages: 21 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Actual)
Dates: Start 2003-06; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Relapse-free survival | Until relapsing

SECONDARY OUTCOMES:
Overall survival | Overall
Local-recurrence-free survival | Until local-recurrence
Incidence of adverse events | 5 years
Incidence of major adverse events | 5 years
Operative time | Operation day
Blood loss | Operation day
Incidence of sexual and urinary dysfunction | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Shin Fujita, MD, Study Chair — National Cancer Center Hospital
Locations (48):
- Japan (48):
  - Aichi Cancer Center Hospital, Nagoya,Chikusa-ku,Kanokoden,1-1, Aichi-ken
  - Fujita Health University, Toyoake,Kutsukake-cho,Dengakugakubo,1-98, Aichi-ken
  - Chiba Cancer Center Hospital, Chiba,Chuo-ku,Nitona-cho,666-2, Chiba
  - National Cancer Center Hospital East, Kashiwa,Kashiwanoha,6-5-1, Chiba
  - Toho University Sakura Hospital, Sakura,Shimoshidu,564-1, Chiba
  - Jyuntendo Urayasu Hospital, Urayasu,Tomioka,2-1-1, Chiba
  - National Hospital Organization Shikoku Cancer Center, Matsuyama,Horinouchi,13, Ehime
  - National Kyushu Cancer Center, Fukuoka,Minami-ku,Notame,3-1-1, Fukuoka
  - Kurume University School of Medicine, Kurume,Asahi-machi,67, Fukuoka
  - Kurume University Medical Center, Kurume,Kokubumachi,155-1, Fukuoka
  - Gunma Prefectural Cancer Center, Ota,Takabayashi-nishi-cho,617-1, Gunma
  - Hiroshima University, School of Medicine, Hiroshima,Minami-ku,Kasumi,1-2-3, Hiroshima
  - Hiroshima City Hospital, Hiroshima,Naka-ku,Motomachi,7-33, Hiroshima
  - Sapporo-Kosei General Hospital, North-3,East8-5,Chuou-ku,Sapporo, Hokkaido
  - Kansai Rosai Hospital, Amagasaki,Inabasou,3-1-69, Hyōgo
  - Ibaraki Kenritsu Chuo Hospital & Cancer Center, Nishi-ibarakigun,Tomobemachi,Koibuchi,6528, Ibaraki
  - Ishikawa Prefectual Central Hospital, Kanazawa,Kuratsuki-Higashi,2-1, Ishikawa-ken
  - Teikyo University Hospital, Mizonokuchi, Kawasaki,Takatsu-ku,Mizonokuchi,3-8-3, Kanagawa
  - Kitasato University East Hospital, Sagamihara,Asamizodai,2-1-1, Kanagawa
  - Kitasato University School of Medichine, Sagamihara,Kitasato,1-15-1, Kanagawa
  - Kanagawa Cancer Center, Yokohama,Asahi-ku,Nakao,1-1-2, Kanagawa
  - Yokohama City University Medical Center, Yokohama,Minami-ku,Urafunecho,4-57, Kanagawa
  - Showa University Northern Yokohama Hospital, Yokohama,Tsuzuki-ku,Chigasakichuo,35-1, Kanagawa
  - National Hospital Organization Kyoto Medical Center, Kyoto,Fushimi-ku,Fukakusa,Mukaihata-cho,1-1, Kyoto
  - Miyagi Cancer Center, Natori,Medeshima-Shiode,Nodayama,47-1, Miyagi
  - Nagano Municipal Hospital, Nagano,Tomitake,1333-1, Nagano
  - Niigata Cancer Center Hospital, Niigata,Kawagishi-cho,2-15-3, Niigata
  - Oita University Fuculty of Medicine, Oita,Hasama-machi,Oogaoka,1-1, Oita Prefecture
  - Okayama Saiseikai General Hospital, Okayama,Ifukucho,1-17-18, Okayama-ken
  - Minoh City Hospital, Minoh,Kayano,5-7-1, Osaka
  - Osaka National Hospital, Osaka,Chuo-ku,Hoenzaka,2-1-14, Osaka
  - Osaka Medical Center for Cancer and Cardiovascular Diseases, Osaka,Higashinari-ku,Nakamichi,1-3-3, Osaka
  - Osaka City General Hospital, Osaka,Miyakojima-ku,Miyakojimahondori,2-13-22, Osaka
  - Sakai Municipal Hospital, Sakai,Minamiyasuicho,1-1-1, Osaka
  - Osaka University Graduate School of Medicine, Suita,Yamada-oka,2-2, Osaka
  - Osaka Medical College, Takatsuki,Daigakucho,2-7, Osaka
  - Omiya Medical Center, Jichi Medical School, Saitama,Omiya-ku,Amanuma-cho,1-847, Saitama
  - National Defense Medical College, Tokorozawa,Namiki,3-2, Saitama
  - Sizuoka Cancer Center, Sunto-gun,Nagaizumi-cho,Shimonagakubo,1007, Shizuoka
  - Tochigi Cancer Center, Utsunomiya,Yohnan,4-9-13, Tochigi
  - Tokyo Medical and Dental University Hospital, Bunkyo-ku,Yushima,1-5-45, Tokyo
  - National Cancer Center Hospital, Chuo-ku,Tsukiji, 5-1-1, Tokyo
  - Toho University Ohashi Hospital, Meguro-ku,Ohashi,2-17-6, Tokyo
  - Toranomon Hospital, Minato-ku,Toranomon,2-2-2, Tokyo
  - Kyorin University School of Medicine, Mitaka,Shinkawa,6-20-2, Tokyo
  - Tokyo Medical University, Shinjuku-ku,Nishi-shinjuku,6-7-1, Tokyo
  - Keio University Hospital, Shinjuku-ku,Shinanomachi,35, Tokyo
  - Yamagata Prefectural Central Hospital, Yamagata,Aoyagi,1800, Yamagata

REFERENCES:
- [Derived] Tsukamoto S, Fujita S, Ota M, Mizusawa J, Shida D, Kanemitsu Y, Ito M, Shiomi A, Komori K, Ohue M, Akazai Y, Shiozawa M, Yamaguchi T, Bando H, Tsuchida A, Okamura S, Akagi Y, Takiguchi N, Saida Y, Akasu T, Moriya Y; Colorectal Cancer Study Group of Japan Clinical Oncology Group. Long-term follow-up of the randomized trial of mesorectal excision with or without lateral lymph node dissection in rectal cancer (JCOG0212). Br J Surg. 2020 Apr;107(5):586-594. doi: 10.1002/bjs.11513. Epub 2020 Mar 12. PMID 32162301
- [Derived] Saito S, Fujita S, Mizusawa J, Kanemitsu Y, Saito N, Kinugasa Y, Akazai Y, Ota M, Ohue M, Komori K, Shiozawa M, Yamaguchi T, Akasu T, Moriya Y; Colorectal Cancer Study Group of Japan Clinical Oncology Group. Male sexual dysfunction after rectal cancer surgery: Results of a randomized trial comparing mesorectal excision with and without lateral lymph node dissection for patients with lower rectal cancer: Japan Clinical Oncology Group Study JCOG0212. Eur J Surg Oncol. 2016 Dec;42(12):1851-1858. doi: 10.1016/j.ejso.2016.07.010. Epub 2016 Jul 30. PMID 27519616
- [Derived] Fujita S, Akasu T, Mizusawa J, Saito N, Kinugasa Y, Kanemitsu Y, Ohue M, Fujii S, Shiozawa M, Yamaguchi T, Moriya Y; Colorectal Cancer Study Group of Japan Clinical Oncology Group. Postoperative morbidity and mortality after mesorectal excision with and without lateral lymph node dissection for clinical stage II or stage III lower rectal cancer (JCOG0212): results from a multicentre, randomised controlled, non-inferiority trial. Lancet Oncol. 2012 Jun;13(6):616-21. doi: 10.1016/S1470-2045(12)70158-4. Epub 2012 May 15. PMID 22591948
- See also: Related Info — http://www.jcog.jp/